CLINICAL TRIAL: NCT02412475
Title: Epigenetic Reprogramming in Relapse AML: A Phase 1 Study of Decitabine and Vorinostat Followed by Fludarabine, Cytarabine and G-CSF (FLAG) in Children and Young Adults With Relapsed/Refractory AML
Brief Title: Epigenetic Reprogramming in Relapse AML
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: We opened a competing study with the TACL consortium
Sponsor: Michael Burke (Other)
Collaborators: Children's Hospitals and Clinics of Minnesota (Other)
Responsible Party: Sponsor-Investigator, Michael Burke, Associate Professor of Pediatrics, Medical College of Wisconsin
Organization: Medical College of Wisconsin (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Epigenetic
Record Dates: First submitted 2015-04-06; First posted 2015-04-09 (Estimated); Last update posted 2019-01-24 (Actual); Status verified 2019-01

CONDITIONS: Leukemia, Acute Myeloid
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Decitabine; Vorinostat; fludarabine; fludarabine phosphate; Cytarabine; Filgrastim; Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment Plan - 2 treatment courses (Experimental): Drug Method Used to Give Drug Days Cytarabine IT 0 or -1 Decitabine IV over 1 hour 1-5 Vorinostat PO 1-5 Fludarabine IV over 30 minutes 6-10 Cytarabine IV over 3 hours 6-10 Filgrastim (G-CSF) IV or SQ 5-12 Sorafenib PO 11-28
  Interventions: Drug: Decitabine; Drug: Vorinostat; Drug: Fludarabine; Drug: Cytarabine; Drug: Filgrastim; Drug: Sorafenib

INTERVENTIONS:
Drug: Decitabine — Dosing per protocol starting at hour 0 IV infusion over 1 hour on Days 1-5
  Other Names: 5-AZA-2'-Deoxycytidine, Dacogen
Drug: Vorinostat — 180 mg per meter squared per day for those under age 18, 300mg BID for those age 18 and older. Given after the decitabine infusion by mouth on Days 1-5
  Other Names: Suberoylanilide Hydroxamic Acid; Zolinza
Drug: Fludarabine — 30 mg per meter squared per day starting at hour 0 given immediately after G-CSF by IV infusion over 30 minutes on days 6-10
  Other Names: Oforta; Fludara
Drug: Cytarabine — 2000 mg per meter squared per day starting at hour 4 by IV over 3 hours on days 6-10
  Other Names: Depocyt
Drug: Filgrastim — 5 μ/kg/dose starting at hour 0 immediately before fludarabine by IV or SQ on days 5-12
  Other Names: Neupogen
Drug: Cytarabine — Patient Age (years) IT Cytarabine Dose > 1 30 mg
  * 2 and < 3 50 mg
  * 3 and ≤ 18 70 mg > 18 100 mg
  given IT on day 0 or -1
  Other Names: Depocyt
Drug: Sorafenib — 150 mg/m2/dose twice daily by mouth on days 11-28
  Other Names: Nexavar

SUMMARY:
Successful treatment for children and young adults with relapsed acute myeloid leukemia (AML) continues to be a significant challenge. Despite relative improvements in survival for patients with newly diagnosed AML, an estimated 40-60% will relapse with the majority eventually dying of their relapsed disease. Attaining a subsequent remission in patients who relapse is the initial critical step toward achieving a potential cure. As chemotherapy resistance is one of the primary drivers of poor treatment response and subsequent relapse in AML, identifying methods to reverse this resistance are desperately needed. This clinical trial is aimed at improving the remission re-Induction rates for children and adults with relapsed or refractory AML through epigenetic modifying agents that have the ability to reverse chemotherapy resistance. Decitabine, a DNA methyltransferase inhibitor (DNMTi) and Vorinostat, a histone deacetylase inhibitor (HDACi), are two epigenetic modifying drugs that act on the methylation of proximal promoter regions of genes and on proteins involved in the wrapping of DNA around histones, respectively. Both processes play a critical role in regulating gene expression, and frequently these genes are involved in chemotherapy resistance. These agents are FDA-approved for treatment in adult hematologic malignancies, making this an opportune time to begin testing these novel therapies in pediatric leukemia trials. This study will investigate chemotherapy priming of relapsed/refractory AML using Decitabine and Vorinostat given for 5 days prior to standard re-Induction with Fludarabine, Cytarabine and G-CSF for children and adults.

DETAILED DESCRIPTION:
Phase 1 Study Number of Patients: 12 to 24 evaluable subjects will be required to enroll subjects in all 4 dose levels.

Study Objectives:

Primary Objectives

* To determine the maximum tolerated dose (MTD) of decitabine when used in this combination with vorinostat, fludarabine, high dose cytarabine and G-CSF (FLAG) for children and young adults with relapsed or refractory AML.
* To evaluate the ability to safely deliver the combination of decitabine and vorinostat followed by fludarabine, high dose cytarabine and G-CSF (FLAG) in pediatric and young adult patients with relapsed or refractory AML.

Secondary Objectives o To establish the extent of hypomethylation of peripheral blood (PB) and bone marrow (BM) pre- and post- decitabine and vorinostat treatment by: LINE-1 methylation assay as a surrogate marker of global DNA methylation. Direct Comprehensive DNA methylation analysis Gene expression profiling to assess genetic changes

* To analyze the correlation between DNA methylation and gene expression pre- and post-treatment with decitabine and vorinostat.
* To analyze the correlation between biological changes and clinical response

Selection of Study Patients:

• Study entry is open to patients regardless of gender or ethnic background. While there will be every effort to seek out and include females and minority patients, the patient population is expected to be no different than that of other acute leukemia studies at the Medical College of Wisconsin.

ELIGIBILITY:
Inclusion Criteria:

The eligibility criteria listed below are interpreted literally and cannot be waived.

• Age: Patients must be ≥ 1 and ≤ 25 years of age when originally diagnosed with AML.

* Diagnosis:

  o Patients must have a diagnosis of AML with > 5% blast in the bone marrow and fall into one of the categories listed below:
* Any patient in 1st or greater relapse OR Patients failed to go into remission after first or greater relapse OR Patients failed to go into remission from original diagnosis after two or more induction attempts.

  o Patients with CNS 1 or CNS 2 leukemia are eligible
* Performance Level: (See Appendix 2 for Performance Scales)

  o Karnofsky Performance Status ≥ 50% for patients 16 years and older

  o Lansky Play Score ≥ 50 for patients under 16 years of age
* Life Expectancy:

  o Patients must have a life expectancy ≥ 8 weeks as determined by the enrolling investigator.
* Prior Therapy:

  o Cytotoxic Therapy: At least 7 days must have elapsed from prior chemotherapy with the exception of hydroxyurea which can be used up to 24 hours of starting this protocol therapy.

  o Hematopoietic Stem Cell Transplant (HSCT): Patients who have experienced their relapse after a HSCT are eligible, provided they have no evidence of active Graft-versus-Host Disease (GVHD).

  o Prior Demethylating and/or HDAC Inhibitor Therapy: Patients who have received prior DNMTi (e.g. decitabine) and/or HDACi (e.g. vorinostat) are eligible to participate in this Phase 1 study.

  o Biologic (anti-neoplastic agent): At least 7 days after the last dose of a biologic agent. For agents that have known adverse events occurring beyond 7 days after administration, this period must be extended beyond the time during which adverse events are known to occur. The duration of this interval must be discussed with the study chair

  o Monoclonal Antibodies: At least 3 half-lives of the antibody must have elapsed after the last dose of monoclonal antibody. (i.e. Gemtuzumab = 36 days)
  * Immunotherapy: At least 42 days after the completion of any type of immunotherapy, e.g. tumor vaccines.
  * XRT: > 14 days for local palliative XRT for CNS chloromas; No washout period is necessary for other chloromas; > 30 days must have elapsed if prior TBI, craniospinal XRT.
* Organ Function:

  * Patients must have acceptable organ function as defined within 7 days of study registration
  * Renal: creatinine clearance ≥ 60 mL/min/1.73 m2 or serum creatinine based on age and gender as follows:

Maximum Serum Creatinine (mg/dL) Age Male Female 1 month to < 6 months 0.4 0.4 6 months to < 1 year 0.5 0.5

1. year to < 2 years 0.6 0.6
2. years to < 6 years 0.8 0.8

6 years to < 10 years 1.0 1.0 10 years to < 13 years 1.2 1.2 13 years to < 16 years 1.5 1.4

* 16 years 1.7 1.4

  * Hepatic: ALT < 5 × upper limit of normal (ULN) and total bilirubin ≤ 1.5 × upper limit of normal (ULN) for age. The hepatic requirements are waived for patients with known or suspected leukemia liver involvement who would otherwise be eligible after consultation with the Study Chair or Vice Chair.
  * Cardiac: left ventricular shortening fraction > 27% by ECHO/MUGA or an ejection fraction ≥ 40% by ECHO/MUGA

    * Reproductive Function:
  * Female patients of childbearing potential must have a negative urine or serum pregnancy test confirmed prior to enrollment.
  * Female patients with infants must agree not to breastfeed their infants while on this study.
  * Male and female patients of child-bearing potential must agree to use an effective method of contraception approved by the investigator during the study.

    • Sexually active females of child bearing potential must agree to use adequate contraception (diaphragm, birth control pills, injections, intrauterine device [IUD], surgical sterilization, subcutaneous implants, or abstinence, etc.) for the duration of treatment and for 2 months after the last dose of chemotherapy. Sexually active men must agree to use barrier contraceptive for the duration of treatment and for 2 months after the last dose of chemotherapy.
    * Voluntary written consent before performance of any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the subject at any time without prejudice to future medical care.

Exclusion Criteria:

Patients will be excluded if they meet any of the following criteria

* They are unable to swallow Vorinostat capsules or take oral solution.
* They are currently receiving other investigational drugs.
* There is a plan to administer non-protocol chemotherapy, radiation therapy, or immunotherapy during the study period.
* They have significant concurrent disease, illness, psychiatric disorder or social issue that would compromise patient safety or compliance, interfere with consent, study participation, follow up, or interpretation of study results.
* They have a known allergy to any of the drugs used in the study.
* Patients with Down syndrome are excluded.
* They are receiving Valproic Acid (VPA) therapy.
* Patients with Acute Promyelocytic Leukemia (APL, APML) are excluded
* Patients with documented active and uncontrolled infection at the time of study entry are not eligible.

Ages: 1 Year to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 3 (Actual)
Dates: Start 2015-02-21 (Actual); Primary Completion 2017-06-21 (Actual); Study Completion 2017-06-21 (Actual)

PRIMARY OUTCOMES:
Achievement of Complete Remission by Bone Marrow Criteria | 60 days
  Complete Remission (CR): Attainment of M1 bone marrow with no evidence of circulating blasts or extramedullary disease and with recovery of peripheral counts (ANC > 750/µL and PLT count > 75,000/µL). Qualifying marrow and peripheral counts should be performed within 1 week of each other. M1 Marrow: Less than 5% blasts in a bone marrow aspirate and at least 200 cells counted

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Burke, MD, Principal Investigator — Medical College of Wisconsin/Children's Hospital of Wisconsin
Locations (2):
- United States (2):
  - Children's Hospitals and Clinics of Minnesota, Minneapolis, Minnesota
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin

REFERENCES:
- [Derived] Pommert L, Schafer ES, Malvar J, Gossai N, Florendo E, Pulakanti K, Heimbruch K, Stelloh C, Chi YY, Sposto R, Rao S, Huynh VT, Brown P, Chang BH, Colace SI, Hermiston ML, Heym K, Hutchinson RJ, Kaplan JA, Mody R, O'Brien TA, Place AE, Shaw PH, Ziegler DS, Wayne A, Bhojwani D, Burke MJ. Decitabine and vorinostat with FLAG chemotherapy in pediatric relapsed/refractory AML: Report from the therapeutic advances in childhood leukemia and lymphoma (TACL) consortium. Am J Hematol. 2022 May;97(5):613-622. doi: 10.1002/ajh.26510. Epub 2022 Mar 8. PMID 35180323